CLINICAL TRIAL: NCT05939193
Title: Effect of Urine-guided Intraoperative Hydration on the Incidence of Postoperative Acute Kidney Injury and Long-term Outcomes in Patients With Pseudomyxoma Peritonei Receiving CRS-HIPEC: a Prospective, Randomized, Controlled Trial
Brief Title: Effect of Urine-guided Hydration on Acute Kidney Injury After CRS-HIPEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Aerospace Center Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anaesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023-080
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cytoreductive Surgery; Hyperthermic Intraperitoneal Chemotherapy; Hydration; Diuresis; Acute Kidney Injury; Postoperative Complications
Keywords: Cytoreductive Surgery; Hyperthermic Intraperitoneal Chemotherapy; Hydration; Diuresis; Acute Kidney Injury; Postoperative Complications
MeSH Terms: conditions — Acute Kidney Injury; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urine-guided hydration (Experimental): The target is to maintain urine output at 200 ml/h (3 ml/kg/h) or higher by intravenous injection/infusion of furosemide throughout surgery. That is, a loading dose of 20 mg is injected at the beginning of surgery; if the urine output does not reach the target value, furosemide will be continuously infused at 10 mg/h until the end of the surgery as needed, with a maximum cumulative dose not exceeding 250 mg. Intravenous hydration is performed to balance urine output and to maintain the SVV≤10%.
  Interventions: Procedure: Urine-guided hydration; Drug: Forced administration of furosemide
- Routine hydration (Active Comparator): The target is to maintain urine output at 0.5 ml/kg/h or higher as per current medical practice. That is, furosemide is only administered when clinically necessary or at the discretion of attending anesthesiologists. Intravenous hydration is performed to maintain the SVV≤10%.
  Interventions: Procedure: Routine hydration; Drug: Routine administration of furosemide

INTERVENTIONS:
Procedure: Urine-guided hydration — The target is to maintain urine output at 200 ml/h (3 ml/kg/h) or higher by intravenous injection/infusion of furosemide throughout surgery. That is, a loading dose of 20 mg is injected at the beginning of surgery; if urine output does not reach the target value, furosemide will be continuously infused at 10 mg/h until the end of surgery, with a cumulative dose not exceeding 250 mg. Intravenous rehydration is performed to balance urine output and to maintain the SVV ≤10%.
  Other Names: Forced administration of furosemide
  Arms: Urine-guided hydration
Procedure: Routine hydration — The target is to maintain urine output at 0.5 ml/kg/h or higher according to routine practice. That is, furosemide is only administered when clinically necessary or at discretion of responsible anesthesiologists; intravenous rehydration is performed to maintain the SVV ≤10%.
  Other Names: Routine administration of furosemide
  Arms: Routine hydration
Drug: Forced administration of furosemide — Forced administration of furosemide
  Arms: Urine-guided hydration
Drug: Routine administration of furosemide — Routine administration of furosemide
  Arms: Routine hydration

SUMMARY:
Acute renal injury (AKI) is a common complication after cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy (CRS-HIPEC), and is associated with worse outcomes. Available evidences show that maintaining intraoperative urine output ≥ 200 ml/h by fluid and furosemide administration may reduce the incidence of AKI in patients undergoing cardiopulmonary bypass. The investigators hypothesize that, for patients undergoing CRS-HIPEC, intraoperative urine-volume guided hydration may also reduce the incidence of postoperative AKI.

DETAILED DESCRIPTION:
Acute renal injury (AKI) is a common complication after cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy (CRS-HIPEC), and is associated with worse outcomes. Studies showed that less intraoperative urine volume was associated with AKI.

In studies of contrast-associated AKI, intraoperative and 4-h postoperative hydration and forced diuresis to achieve urine output ≥ 300 ml/h reduces the incidence of AKI by 44%. In patients undergoing cardiac surgery under cardiopulmonary bypass, maintaining intraoperative and 6-h postoperative urine output ≥200 ml/h by fluid and furosemide administration reduces the incidence of AKI by 52%. For patients with rhabdomyolysis, it is recommended to maintain urine output at approximately 3 ml/kg/h (200 ml/h) with volume supplementation. We suppose that forced diuresis with simultaneous hydration (balancing urine output with intravenous fluid infusion) may reduce AKI after CRS-HIPEC.

The purpose of this randomised controlled trial is to investigate whether maintaining urine output at 200 ml/h (3 ml/kg/h) or higher by forced diuresis with simultaneous hydration can reduce the incidence of AKI after CRS-HIPEC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosed as pseudomyxoma peritonei, scheduled for cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy under general anesthesia;
* At least 14 days since the last treatment of chemotherapy, radiotherapy, or immunotherapy;
* Consent to participate in this study.

Exclusion Criteria:

* Persistent preoperative atrial fibrillation, or new-onset cardiovascular event (acute coronary syndrome, stroke, or congestive heart failure) in the past 3 months;
* Requirement of vasopressors to maintain blood pressure before surgery;
* Known furosemide hypersensitivity;
* Chronic kidney disease stage 5 or requirement of renal replacement therapy;
* Other conditions that are considered unsuitable for the study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury (AKI) within 7 days after surgery | Up to 7 days after surgery
  Acute kidney injury (AKI) is diagnosed according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria.

SECONDARY OUTCOMES:
Classification of AKI within 7 days after surgery | Up to 7 days after surgery
  AKI is classified according to the KDIGO criteria.
Intensive care unit (ICU) admission after surgery | Up to 30 days after surgery
  ICU admission after surgery
Length of ICU stay after surgery | Up to 30 days after surgery
  Length of ICU stay after surgery
Duration of mechanical ventilation after surgery | Up to 30 days after surgery
  Duration of mechanical ventilation after surgery
Length of hospital stay after surgery | Up to 30 days after surgery
  Length of hospital stay after surgery
Incidence of other organ injuries within 7 days after surgery | Up to 7 days after surgery
  Including delirium (assessed with the Confusion Assessment Method [3D-CAM] for patients without mechanical ventilation and CAM-ICU for patients with mechanical ventilation]) within 5 days after surgery, myocardial injury and other organ injuries other than AKI.
All-cause 30-day mortality | Up to 30 days after surgery
  All-cause 30-day mortality
Incidence of postoperative major complications | Up to 30 days after surgery
  Postoperative major complications were defined as new-onset conditions that were harmful for patients' recovery and required therapeutic intervention, i.e., grade 2 or higher on Clavien-Dindo classification.

OTHER OUTCOMES:
Incidence of deterioration in renal function | Up to 6 months after surgery
  Defined as ≥1 grade decrease in glomerular filtration rate compared with preoperative value.
Recurrence/progress-free survival | Up to 6 months after surgery
  Defined as time from surgery to pseudomyxoma peritonei recurrence/progress/metastasis or all-cause death, whichever occurs first.
Event-free survival | Up to 6 months after surgery
  Defined as time from surgery to pseudomyxoma peritonei recurrence/progress/metastasis, unplanned re-hospitalization for non-pseudomyxoma peritonei diseases, or all-cause death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital, Beijing, CHINA
Locations (1):
- Aerospace Center Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liesenfeld LF, Wagner B, Hillebrecht HC, Brune M, Eckert C, Klose J, Schmidt T, Buchler MW, Schneider M. HIPEC-Induced Acute Kidney Injury: A Retrospective Clinical Study and Preclinical Model. Ann Surg Oncol. 2022 Jan;29(1):139-151. doi: 10.1245/s10434-021-10376-5. Epub 2021 Jul 14. PMID 34260006
- [Background] Angeles MA, Quenet F, Vieille P, Gladieff L, Ruiz J, Picard M, Migliorelli F, Chaltiel L, Martinez-Gomez C, Martinez A, Ferron G. Predictive risk factors of acute kidney injury after cytoreductive surgery and cisplatin-based hyperthermic intra-peritoneal chemotherapy for ovarian peritoneal carcinomatosis. Int J Gynecol Cancer. 2019 Feb;29(2):382-391. doi: 10.1136/ijgc-2018-000099. Epub 2019 Jan 23. PMID 30674567
- [Background] Hakeam HA, Breakiet M, Azzam A, Nadeem A, Amin T. The incidence of cisplatin nephrotoxicity post hyperthermic intraperitoneal chemotherapy (HIPEC) and cytoreductive surgery. Ren Fail. 2014 Nov;36(10):1486-91. doi: 10.3109/0886022X.2014.949758. Epub 2014 Aug 26. PMID 25155314
- [Background] Markowiak T, Kerner N, Neu R, Potzger T, Grosser C, Zeman F, Hofmann HS, Ried M. Adequate nephroprotection reduces renal complications after hyperthermic intrathoracic chemotherapy. J Surg Oncol. 2019 Dec;120(7):1220-1226. doi: 10.1002/jso.25726. Epub 2019 Oct 10. PMID 31602673
- [Background] Solanki SL, Mukherjee S, Agarwal V, Thota RS, Balakrishnan K, Shah SB, Desai N, Garg R, Ambulkar RP, Bhorkar NM, Patro V, Sinukumar S, Venketeswaran MV, Joshi MP, Chikkalingegowda RH, Gottumukkala V, Owusu-Agyemang P, Saklani AP, Mehta SS, Seshadri RA, Bell JC, Bhatnagar S, Divatia JV. Society of Onco-Anaesthesia and Perioperative Care consensus guidelines for perioperative management of patients for cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (CRS-HIPEC). Indian J Anaesth. 2019 Dec;63(12):972-987. doi: 10.4103/ija.IJA_765_19. Epub 2019 Dec 11. PMID 31879421
- [Background] Briguori C, D'Amore C, De Micco F, Signore N, Esposito G, Visconti G, Airoldi F, Signoriello G, Focaccio A. Left Ventricular End-Diastolic Pressure Versus Urine Flow Rate-Guided Hydration in Preventing Contrast-Associated Acute Kidney Injury. JACC Cardiovasc Interv. 2020 Sep 14;13(17):2065-2074. doi: 10.1016/j.jcin.2020.04.051. PMID 32912462
- [Background] Luckraz H, Giri R, Wrigley B, Nagarajan K, Senanayake E, Sharman E, Beare L, Nevill A. Reduction in acute kidney injury post cardiac surgery using balanced forced diuresis: a randomized, controlled trial. Eur J Cardiothorac Surg. 2021 Apr 13;59(3):562-569. doi: 10.1093/ejcts/ezaa395. PMID 33236105
- [Background] Bosch X, Poch E, Grau JM. Rhabdomyolysis and acute kidney injury. N Engl J Med. 2009 Jul 2;361(1):62-72. doi: 10.1056/NEJMra0801327. No abstract available. PMID 19571284